CLINICAL TRIAL: NCT04482257
Title: *Official Title: Randomized, Open-label, Single-dose, Two-sequence, Two-period, Crossover Bioequivalence Trial of Irinotecan Liposome Injection in Patients With Advanced Pancreatic Cancer.
Brief Title: Bioequivalence Study of Irinotecan Liposome Injection in Chinese Advanced Pancreatic Cancer.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HE072-BE-002
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Advanced Pancreatic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-R (Experimental): Subjects will receive Irinotecan Liposome Injection (CSPC) 70mg/m2 plus 5-FU/LV, followed by Irinotecan Liposome Injection (Ipsen) 70mg/m2 plus 5-FU/LV
  Interventions: Drug: Irinotecan Liposome Injection combined with 5-FU/LV
- R-T (Experimental): Subjects will receive Irinotecan Liposome Injection (Ipsen) 70mg/m2 plus 5-FU/LV, followed by Irinotecan Liposome Injection (CSPC) 70mg/m2 plus 5-FU/LV
  Interventions: Drug: Irinotecan Liposome Injection combined with 5-FU/LV

INTERVENTIONS:
Drug: Irinotecan Liposome Injection combined with 5-FU/LV — Drug: Irinotecan Liposome Injection 70mg/m2 (CSPC) combined with 5-FU/LV; Drug: Irinotecan Liposome Injection 70mg/m2 (Ipsen, ONIVYDETM) combined with 5-FU/LV;

SUMMARY:
Randomized, Open-label, Single-dose, Two-sequence, Two-period, Crossover Bioequivalence Trial of Irinotecan Liposome Injection in Patients With Advanced Pancreatic Cancer.

DETAILED DESCRIPTION:
The purpose of this study was to determine the bioequivalence of two formulations of Irinotecan Liposome Injection (70mg/m2) in Chinese patients with Advanced Pancreatic Cancer, under fasting condition. These data were to be evaluated statistically to determine if the products meet bioequivalence criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent for participation in the trial.
2. Advanced pancreatic cancer diagnosed by histopathology and / or cytology.
3. Age ≥ 18 years, men or women. BMI is above 17.
4. ECOG score 0 to 2.
5. Life expectancy ≥ 3 months.
6. Adequate bone marrow function.
7. Adequate hepatic function.
8. Adequate renal function.
9. Patient with reproductive potential must agree to use adequate contraception from the signing of informed consent to at least 6 months after the trial

Exclusion Criteria:

1. Patients who have a severe allergy or a significant history of hypersensitivity or an idiopathic reaction attributed to irinotecan or compounds of similar chemical composition to irinotecan ;
2. Patients who have previously used irinotecan liposomes and experienced treatment failure or serious adverse reactions;
3. Patients with severe cardiovascular, lung, liver, kidney, gastrointestinal, endocrine, immune system, skin, musculoskeletal, neurological or psychiatric diseases that occurred within 3 months of the first dose of the study drug, and not suitable for this study as determined by the researchers;
4. Patients who have undergone major surgery within 4 weeks of screening or have a schedule for major surgery during the study period;
5. Patients who have received any radiotherapy or chemotherapy and other anti-tumor treatment within 4 weeks of the first dose of the study drug, traditional Chinese medicine with anti-tumor indications within 4 weeks of the first dose of the study drug, or small molecule targeted drugs within 2 weeks (or 5 half-lives whichever is longer) of the first dose of the study drug;
6. Patients who currently enrolled in any other clinical study, or received other investigational agents within 4 weeks of the first dose of the study drug；
7. Blood donation or massive blood loss (>400mL) within 90 days of screening;
8. Concomitant use of strong CYP3A4 inhibitors or inducers, or UGT1A1 inhibitors within 4 weeks of the first dose of the study drug;
9. Patients who received certain diet (such as grapefruit) which may interfere with the evaluation of PK results;
10. LVEF≤50%;
11. Patients with extended QT/QTc interval (QTcF>480ms);
12. History of alcohol or drugs abuse;
13. Pregnant or lactating women;
14. Patients with known Hepatitis B Virus (HBV DNA≥104), Hepatitis C Virus (anti-HCV positive, HCV RNA positive), Human immunodeficiency virus antibody (anti-HIV positive), or active Treponema Pallidum viral infection;
15. Patients with homozygous UGT1A1*28 genotype or UGT1A1*6 genotype;
16. Patients who are not suitable for this study as determined by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Cmax | 0 -190 hours
  Cmax of Total Irinotecan and Free Irinotecan will be measured for the test product (CSPC) or the reference product (Ipsen).
AUC0-t | 0 -190 hours
  The exposure of Total Irinotecan and Free Irinotecan from time (0) to the last quantifiable concentration (t) will be measured for the test product (CSPC) or the reference product (Ipsen).
AUC0-∞ | 0 -190 hours
  The exposure of Total Irinotecan and Free Irinotecan from time (0) to infinity (∞) will be calculated for the test product (CSPC) or the reference product (Ipsen).
Tmax | 0 -190 hours
  The time to maximum concentration will be measured for the test product (CSPC) or the reference product (Ipsen).
t1/2 | 0 -190 hours
  The terminal elimination half-life will be calculated for the test product (CSPC) or the reference product (Ipsen).
λz | 0 -190 hours
  The terminal elimination rate constant will be calculated for the test product (CSPC) or the reference product (Ipsen).

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, Ph.D, Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No